CLINICAL TRIAL: NCT05203237
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VK2735, a Dual Glucagon-like Peptide-1 and Gastric Inhibitory Polypeptide Receptor Agonist, in Healthy Adults and Otherwise Healthy Adults Who Have an Increased Body Mass Index
Brief Title: Phase 1 Study to Evaluate the Safety and Tolerability of VK2735
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VK2735-101
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Weight Loss; NASH
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Part A) (Placebo Comparator): Placebo administered SC once in healthy participants
  Interventions: Biological: Placebo
- VK2735 (Part A) (Experimental): Escalating doses of VK2735 administered subcutaneously (SC) once in healthy participants.
  Interventions: Biological: VK2735
- Placebo (Part B) (Placebo Comparator): Placebo administered SC once weekly for four weeks in healthy participants
  Interventions: Biological: Placebo
- VK2735 (Part B) (Experimental): Escalating doses of VK2735 administered subcutaneously (SC) once weekly in healthy participants.
  Interventions: Biological: VK2735
- VK2735 (Part C ) (Placebo Comparator): Placebo administered orally daily for 28 days in healthy participants
  Interventions: Drug: VK2735 Placebo
- VK2735 (Part C) (Experimental): Escalating doses of VK2735 administered daily (PO) in healthy participants.
  Interventions: Drug: VK2735 Drug

INTERVENTIONS:
Biological: VK2735 — Administered SC
  Arms: VK2735 (Part A); VK2735 (Part B)
Biological: Placebo — Administered SC
  Arms: Placebo (Part A); Placebo (Part B)
Drug: VK2735 Placebo — Administered orally
  Arms: VK2735 (Part C )
Drug: VK2735 Drug — Administered orally
  Arms: VK2735 (Part C)

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled single and multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of VK2735 in healthy adults and otherwise healthy adults who have an increased body mass index (BMI).

DETAILED DESCRIPTION:
This study comprises 3 parts:

Part A (Single Ascending Dose [SAD]) will be conducted to assess the safety, tolerability, and PK profile in healthy participants following 1 single SC injection of VK2735 or VK2735 matching placebo (SAD Cohort 1 through SAD Cohort 6).

Part B (Multiple Ascending Dose [MAD]) will be conducted to assess the safety, tolerability, PK and PD profile in otherwise healthy participants who have an increased BMI following single SC injections of VK2735 or matched placebo administered once weekly for 4 consecutive weeks (MAD Cohort 1 through MAD Cohort 5).

Part C (Multiple Ascending Dose [MAD], PO) will be conducted to assess the safety, tolerability, PK and PD profiles in otherwise healthy, but obese, participants who have a BMI ≥30 kg/m2 following daily oral administration of VK2735 or matched placebo administered for 28 consecutive days (MAD-PO Cohort 1 through MAD-PO Cohort 4, with optional additional cohorts)

Safety Review Committee (SRC) meetings will be held prior to dose escalation for Part A (SAD), Part B (MAD), and Part C (MAD-PO) cohorts in the study. The decisions on dose escalation will be based on safety and laboratory data from each cohort.

ELIGIBILITY:
Inclusion Criteria:

Participants must be capable of giving signed informed consent

Participants must be medically healthy, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening and/or before administration of the initial dose of IP in the opinion of the Investigator

Participant body weight must have been stable (no change greater than 5%) for a minimum 8 weeks prior to Screening

Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other clinical study procedures

Willing to comply with contraception requirements

Exclusion Criteria:

Participants with any level of disease or organ system dysfunction as identified during physical examination, medical history or laboratory testing, as assessed by the PI

Any surgical or medical condition (active or chronic) that may interfere with IP distribution, metabolism, excretion, or drug absorption

Participants may be excluded from the study if they have conditions that might compromise safety or other endpoints in the study as judged by the Sponsor (or designee) or Investigator

History or presence of clinically significant acute or unstable cerebrovascular (stroke), hepatic, renal, gastrointestinal, pulmonary, immunological, endocrine, diabetes, hematological, oncological, or central nervous disorder that in the opinion of the Investigator would pose a significant risk for the participant

Use of any investigational drug or product, or participation in an investigational drug study within 30 days prior to dosing or 5 half-lives of the drug (whichever is longest)

Active smoker and/or user of nicotine-containing products unless the participant agrees to discontinue smoking/use of nicotine-containing products from 2 weeks before first IP dose administration through to study completion, including the Follow-up period

Have serum triglycerides > 5.65 mmol/L (500 mg/dL) at Screening

Positive serology for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or HIV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and treatment-emergent serious AEs (TESAEs) | 8 days
  To evaluate the safety and tolerability of single doses of subcutaneous injections of VK2735 in healthy participants

SECONDARY OUTCOMES:
Evaluate the Pharmacokinetic profile of VK2735 | 29 days
  Pharmacokinetic profile of VK2735 by measuring peak plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Mancini, Study Director — Viking Therapeutics, Inc.
Locations (1):
- Viking Clinical Site, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No